CLINICAL TRIAL: NCT06849258
Title: A Prospective, Multicenter, Double Blind, Randomized, Clinical Study to Evaluate the Safety and Efficacy of The FloStent in Men Suffering From Benign Prostatic Hyperplasia Symptoms
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of the FloStent in Men With Benign Prostatic Hyperplasia Symptoms
Acronym: RAPID-III
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rivermark Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C0002 Rev. 07
Record Dates: First submitted 2025-02-17; First posted 2025-02-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia; FloStent; Rivermark Medical; BPH; LUTS; Lower urinary tract symptoms; enlarged prostate
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 2:1 (device:sham) ratio .
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment - FloStent (Experimental): Flexible cystoscopy procedure with FloStent implant deployed
  Interventions: Device: FloStent
- Sham Control (Sham Comparator): Flexible cystoscopy procedure without FloStent implant deployed
  Interventions: Device: Sham (Control)

INTERVENTIONS:
Device: FloStent — Flexible cystoscopy to deploy medical device used to treat BPH
  Arms: Treatment - FloStent
Device: Sham (Control) — Flexible Cystoscopy without deployment of medical device used to treat BPH
  Arms: Sham Control

SUMMARY:
The goal of this study is to determine the safety and effectiveness of the FloStent, a medical device used to treat men with symptoms of Benign Prostatic Hyperplasia, compared to sham (procedure without deployment of the FloStent). All participants will undergo a flexible cystoscopy and those randomized to the treatment arm will receive the FloStent, while those randomized to the sham arm will not receive the FloStent.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects > 45 years of age who have symptomatic BPH
* International Prostate Symptom Score (IPSS) score >13
* Peak urinary flow rate (Qmax): >5 mL/sec and <13 mL/sec with minimum voided volume of >125 mL
* Post-void residual (PVR) <250 mL
* Prostate volume 25 to 80 mL
* Prostatic urethral length 20-50 mm
* Able to complete the study protocol and visits

Exclusion Criteria:

* Presence of an artificial urinary sphincter or stent(s) in the urethra or prostate
* Prior minimally invasive intervention or surgical intervention of the prostate or urethra
* PSA >10 ng/mL
* Bladder cancer or bladder stones
* Active urinary tract infection (UTI)
* Uncontrolled diabetes
* Part of a vulnerable population (cognitively challenged or are incarcerated)

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male at birth and identify as male
Enrollment: 215 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | 12 months
  The International Prostate Symptom Score IPSS is a self-questionnaire (patient reported outcome). It contains 7 questions about symptoms related to BPH and 1 question about the patient's perceived quality of life (QoL).
  The 7 questions are scored from 0 to 5. The sum of the 7 items gives the International Prostate Symptom Score in terms of severity (out of 35):
  0-7 mildly symptomatic 8-19 moderately symptomatic 20-35 severely symptomatic

SECONDARY OUTCOMES:
Percent responders to IPSS | 3 months
  A responder is defined as a subject who has an IPSS improvement ≥ 30% post-treatment as compared to baseline.
Percent responders to IPSS | 6 months
  A responder is defined as a subject who has an IPSS improvement ≥ 30% post-treatment as compared to baseline.
Percent responders to IPSS | 12 months
  A responder is defined as a subject who has an IPSS improvement ≥ 30% post-treatment as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, MD, Study Director — Rivermark Medical, Inc.
Locations (20):
- United States (19):
  - Michael G Oefelein Clinical Trials, Bakersfield, California
  - Comprehensive Urology Medical Group, Beverly Hills, California
  - Atlas Men's Health, La Mesa, California
  - Urology Group of Southern California, Los Angeles, California
  - Prestige Medical Group, Tustin, California
  - Urology Denver, Littleton, Colorado
  - Advanced Urology Institute, Daytona Beach, Florida
  - Duly Health, Lisle, Illinois
  - Loyola Medicine, Maywood, Illinois
  - Southern Urology, Lafayette, Louisiana
  - Michigan Institute of Urology, Troy, Michigan
  - Sheldon Freedman Urology, Las Vegas, Nevada
  - Manhattan Medical Research NYU Langone, New York, New York
  - Northwell Health, Syosset, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Conrad Pearson Clinic, Germantown, Tennessee
  - Midtown Urology Associates, Austin, Texas
  - Urology Austin/Urology America, Austin, Texas
  - Houston Methodist, Houston, Texas
- South Coast Urology, Wollongong, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No